CLINICAL TRIAL: NCT03322137
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2b, Multicenter Study to Evaluate the Safety, Efficacy, and Tolerability of SNA-120 (Pegcantratinib) Ointment in Subjects With Pruritus Associated With Psoriasis Vulgaris
Brief Title: Safety, Efficacy, and Tolerability of SNA-120 in Subjects With Pruritus Associated With Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sienna Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Sienna Labs (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNA-120-201
Record Dates: First submitted 2017-10-04; First posted 2017-10-26 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Pruritus; Psoriasis Vulgaris
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SNA-120 (0.05% ) (Active Comparator): Pegcantratinib Ointment
  Interventions: Drug: SNA-120
- SNA-120 (0.5%) (Active Comparator): Pegcantratinib Ointment
  Interventions: Drug: SNA-120
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: SNA-120 — Pegcantratinib ointment
  Arms: SNA-120 (0.05% ); SNA-120 (0.5%)
Drug: Vehicle — Placebo ointment to mimic Pegcantratinib ointment
  Arms: Vehicle

SUMMARY:
To characterize the efficacy, safety and tolerability of SNA-120 at 2 doses versus placebo when administered topically for the treatment of pruritus associated with psoriasis vulgaris (PV) and PV itself.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent and Health Insurance Portability and Accountability Act (HIPAA) authorization
* Stable PV for at least 6 months prior to screening
* Chronic pruritus of the PV plaques to be present for at least 6 weeks prior to screening
* Mild to moderate PV at screening and baseline
* Has a target plaque at baseline on the trunk and/or limbs
* Subject's plaques are amenable to treatment with a topical ointment medication
* Willing and able to comply with the study instructions and attend all scheduled study visits.
* Willing to avoid prolonged exposure of the designated treatment plaques to ultraviolet radiation
* Females of childbearing potential must have a negative pregnancy test at baseline before randomization and must agree to use highly effective contraception during the study
* Men who are sexually active and can father children must agree to use highly effective forms of contraception during the study

Exclusion Criteria:

* Underlying conditions other than psoriasis that, in the opinion of the investigator, currently cause or influence pruritus of the overall skin
* Positive hepatitis serology
* Thyroid abnormalities that may impact itching
* Subjects with spontaneously improving or rapidly deteriorating PV and/or pruritus
* Current diagnosis of guttate, erythrodermic, exfoliative, or pustular psoriasis
* Active psoriasis or itch affecting the palmar/plantar regions
* Subjects with a clinical diagnosis of bacterial infection of the skin
* Any major medical illness or symptoms of a clinically significant illness that may influence the study outcome
* Any acute chronic medical or psychiatric condition or laboratory abnormality that would make them unsuitable for participation in this study
* Known hypersensitivity to the study treatment excipients and /or polyethylene glycol, that contraindicates participation
* Currently enrolled in an investigational drug or device study or has used an investigational drug or an investigational device treatment within 30 days of randomization/baseline (Note: Subjects who are enrolled in a long-term follow-up study and are not actively receiving an investigational drug or investigational device treatment may be eligible for participation in this study)
* Female who is pregnant or lactating, or is planning to become pregnant during the study
* Subjects participating in any previous SNA-120 (and/or CT327) clinical studies

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Change in Itch Numeric Rating Scale scores (I-NRS) | week 1
  The I-NRS is a 11 point scale, where "0" represents no itch and "10" represents worst possible itching
Change in Itch Numeric Rating Scale scores (I-NRS) | week 2
  The I-NRS is a 11 point scale, where "0" represents no itch and "10" represents worst possible itching
Change in Itch Numeric Rating Scale scores (I-NRS) | week 4
  The I-NRS is a 11 point scale, where "0" represents no itch and "10" represents worst possible itching
Change in Itch Numeric Rating Scale scores (I-NRS) | week 6
  The I-NRS is a 11 point scale, where "0" represents no itch and "10" represents worst possible itching
Change in Itch Numeric Rating Scale scores (I-NRS) | week 8
  The I-NRS is a 11 point scale, where "0" represents no itch and "10" represents worst possible itching

SECONDARY OUTCOMES:
Proportion of subjects (≥ 1 grade change) on IGA scale | week 12
  Investigator Global Assessment
Proportion of subjects (≥ 2 grade change) on IGA scale | week 12
  Investigator Global Assessment
Proportion of subjects categorized as a "0" or "1" on IGA scale and minimum improvement of 2 categories | baseline and week 12
  Investigator Global Assessment
Change in PASI-50 | baseline and week 12
  Percentage of subjects with 50% reductions in Psoriasis Area and Severity Index

OTHER OUTCOMES:
Safety measured by incidence and severity of adverse events | up to 12 weeks
Safety measured by change in clinical laboratory results from baseline | up to 12 weeks
  urinalysis lab assessments
Safety measured by change in clinical laboratory results from baseline | up to 12 weeks
  biochemistry lab assessments
Safety measured by change in clinical laboratory results from baseline | up to 12 weeks
  hematology lab assessments
Safety measured by change in blood pressure from baseline | up to 12 weeks
  systolic/diastolic blood pressure (BP in mmHg)
Safety measured by change in pulse from baseline | up to 12 weeks
  Pulse (beats per minute [bpm])
Safety measured by number of abnormal physical examination changes | baseline and week 12
  Any abnormal physical examination changes from baseline and week 12
Safety measured by PR/PQ intervals measured by 12-lead ECG | week 2
Safety measured by PR/PQ intervals measured by 12-lead ECG | week 8
Safety measured by PR/PQ intervals measured by 12-lead ECG | week 12
Safety measured by QRS duration measured by 12-lead ECG | week 2
Safety measured by QRS duration measured by 12-lead ECG | week 8
Safety measured by QRS duration measured by 12-lead ECG | week 12
Safety measured by QT interval measure by 12-lead ECG | week 2
Safety measured by QT interval measure by 12-lead ECG | week 8
Safety measured by QT interval measure by 12-lead ECG | week 12

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - Site 025, Scottsdale, Arizona
  - Sienna 022, Fort Smith, Arkansas
  - Site 028, Fountain Valley, California
  - Sienna 009, Fremont, California
  - Sienna 008, San Diego, California
  - Sienna 020, Santa Monica, California
  - Sienna 015, Denver, Colorado
  - Sienna 005, Farmington, Connecticut
  - Site 030, Shelton, Connecticut
  - Site 026, Doral, Florida
  - Sienna 019, Largo, Florida
  - Sienna 017, North Miami Beach, Florida
  - Sienna 024, Ocala, Florida
  - Site 027, West Palm Beach, Florida
  - Site 029, Macon, Georgia
  - Sienna 010, New Albany, Indiana
  - Sienna 011, Plainfield, Indiana
  - Sienna 023, Louisville, Kentucky
  - Site 038, Metairie, Louisiana
  - Site 032, Rockville, Maryland
  - Site 039, Clarkston, Michigan
  - Sienna 002, Fridley, Minnesota
  - Sienna 001, St Louis, Missouri
  - Sienna 004, East Windsor, New Jersey
  - Sienna 013, Albuquerque, New Mexico
  - Site 037, Rochester, New York
  - Sienna 016, High Point, North Carolina
  - Sienna 006, Winston-Salem, North Carolina
  - Site 041, Norman, Oklahoma
  - Sienna 003, Portland, Oregon
  - Site 031, Pittsburgh, Pennsylvania
  - Site 035, Murfreesboro, Tennessee
  - Sienna 012, Austin, Texas
  - Sienna 021, Dallas, Texas
  - Sienna 018, Houston, Texas
  - Site 034, Pflugerville, Texas
  - Sienna 007, Murray, Utah
  - Sienna 014, Norfolk, Virginia